CLINICAL TRIAL: NCT05813795
Title: A Phase 3, Multi-center, Randomized, Double-Blind and Placebo-controlled Study to Evaluate the Efficacy and Safety of XW003 in Adults With Overweight or Obesity (SLIMMER)
Brief Title: A Phase 3 Study to Evaluate the Efficacy of XW003 in Adults With Overweight or Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Sciwind Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCW0502-1131
Record Dates: First submitted 2023-03-20; First posted 2023-04-14 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-07

CONDITIONS: Weight Management
Keywords: Weight management; overweight; obesity; glucagon-like peptide-1 (GLP-1); ecnoglutide; XW003
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- C1- XW003 Low Dosage (Experimental): XW003 with low dosage once weekly
  Interventions: Drug: Ecnoglutide Low Dosage
- C1-Placebo (Placebo Comparator): Matched Placebo once weekly
  Interventions: Drug: Placebo
- C2- XW003 Medium Dosage (Experimental): XW003 with medium dosage once weekly
  Interventions: Drug: Ecnoglutide Medium Dosage
- C2-Placebo (Placebo Comparator): Matched Placebo once weekly
  Interventions: Drug: Placebo
- C3- XW003 High Dosage (Experimental): XW003 with high dosage once weekly
  Interventions: Drug: Ecnoglutide High Dosage
- C3-Placebo (Placebo Comparator): Matched Placebo once weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ecnoglutide Low Dosage — Subcutaneous Injection
  Other Names: XW003
  Arms: C1- XW003 Low Dosage
Drug: Ecnoglutide Medium Dosage — Subcutaneous Injection
  Other Names: XW003
  Arms: C2- XW003 Medium Dosage
Drug: Ecnoglutide High Dosage — Subcutaneous Injection
  Other Names: XW003
  Arms: C3- XW003 High Dosage
Drug: Placebo — Subcutaneous Injection with matched volume
  Arms: C1-Placebo; C2-Placebo; C3-Placebo

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of XW003 versus placebo in adults with overweight or obesity

DETAILED DESCRIPTION:
In this Phase 3 study, eligible participants will be randomized into three cohorts in a 3:1:3:1:3:1 ratio to receive once-weekly subcutaneous XW003 (low, medium, or high dosage) or volume-matching placebo for 48 weeks, including a dose-escalation period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-75 years old, inclusive;
2. BMI between 24.0 to 28.0 kg/m2 with at least one comorbidity, including prediabetes, hypertension, hyperlipidemia, fatty liver , obstructive sleep apnea syndrome, etc.; or BMI ≥ 28 kg/m2 with or without comorbidities.
3. Weight change of no more than 5% (based on self-report), with diet and exercise alone, within 3 months before screening.
4. Willing and able to maintain stable diet and exercise during the study period.

Exclusion Criteria:

1. Obesity induced by endocrine diseases such as hypothyroidism, Cushing Syndrome, etc.
2. History of bariatric surgery (except liposuction >1 year ago) or planned bariatric surgery during the study period.
3. Within 3 months before screening, history of using the following drugs or treatments:

   1. Any approved or unapproved weight-loss drugs or Chinese herbs or health products that affect body weight.
   2. Any hypoglycemic medication.
   3. Any medication that may cause significant weight gain, including systemic glucocorticoid treatment, tricyclic anti-depressants, anti-epileptic and antipsychotics.
   4. Any investigational drug, vaccine, or medical device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Percent change in body weight from baseline | Week 40
Proportion of subjects with weight loss ≥5% from baseline | Week 40

SECONDARY OUTCOMES:
Percent and absolute body weight change from baseline | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 32, Week 40 and Week 48
Proportion of subjects with weight loss ≥ 5%, 10%, 15% from baseline | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 32, Week 40 and Week 48
Change from baseline in BMI | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 32, Week 40 and Week 48
  height will be only measured at baseline
Change from baseline in waist and hip circumferences | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 32, Week 40 and Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Dr, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji L, Gao L, Xue H, Tian J, Wang K, Jiang H, Huang C, Lian Q, Yuan M, Gao G, Lu Y, Han J, Fu W, Wang H, Zhang Y, Shi X, Wen B, Shi B, Hu W, Guo T, Xing Y, Li Y, Li Q, Zheng Q, Yang M, Ning J, Guo M, Li Y, Pan H. Efficacy and safety of a biased GLP-1 receptor agonist ecnoglutide in adults with overweight or obesity: a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Diabetes Endocrinol. 2025 Sep;13(9):777-789. doi: 10.1016/S2213-8587(25)00141-X. Epub 2025 Jun 21. PMID 40555243